CLINICAL TRIAL: NCT07021508
Title: Efficacy and Safety Assessment of Temporal Interference Stimulation to Improve Bipolar Depression: a Randomized Controlled Study
Brief Title: Efficacy and Safety Assessment of Temporal Interference Stimulation to Improve Bipolar Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT20250009C-R1
Record Dates: First submitted 2025-05-19; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-02

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temporal Interference Stimulation (Active Comparator)
  Interventions: Device: Temporal Interference Stimulation
- Sham Temporal Interference Stimulation (Sham Comparator)
  Interventions: Device: Sham Temporal Interference Stimulation

INTERVENTIONS:
Device: Temporal Interference Stimulation — A non-invasive, non-invasive method of deep brain electrical stimulation utilizing high-frequency electric field interactions to produce a low-frequency envelope to modulate neural activity.
  Arms: Temporal Interference Stimulation
Device: Sham Temporal Interference Stimulation — The same machine was used as the temporal Interferenc real stimulus, with current creep only 20 seconds before stimulus onset to simulate the real stimulus sensation.
  Arms: Sham Temporal Interference Stimulation

SUMMARY:
The aim of this study was to explore the efficacy and safety of temporal interference stimulation to improve bipolar depression, as well as to explore the corresponding neuroimaging mechanisms using magnetic resonance and electroencephalogram to provide novel intervention protocols and objective indicators of efficacy prediction for depressive episodes in bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* right-handed, and have completed nine years of compulsory education;
* Meet the diagnostic criteria for bipolar depression in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5);
* ≥18 points on the Hamilton Depression Inventory (HAMD- 17);
* ≤8 points on the Young's Mania Rating Scale (YMRS);
* Subjects who have not been treated with psychiatric medication, or those who have been treated with medication are required to undergo medication washout within 2 weeks before randomization;
* Subjects/legal guardians are willing to cooperate with the treatment and sign an informed consent form after they have fully understood the Temporal Interference Stimulation (TI).

Exclusion Criteria:

* Contraindications to magnetic resonance scanning (MRI) or time-interference stimulation (TI), such as the presence of metallic or electronic devices in the body (intracranial metallic foreign bodies, cochlear implants, pacemakers and stents, and other metallic foreign bodies);
* Prior or current electroconvulsive therapy (ECT), modified electroconvulsive therapy (MECT), transcranial magnetic stimulation (TMS), transcranial direct current therapy (tDCS), transcranial alternating current stimulation (tACS), or other neurostimulation;
* Pregnant and lactating women, and women of childbearing age with a positive urine pregnancy;
* Possesses a diagnosis of another major psychiatric disorder that has been assessed by the study investigator as a major disorder that results in more impairment than a diagnosis of bipolar disorder;
* Co-morbid other psychiatric disorders, including obsessive-compulsive disorder, personality disorders, anxiety spectrum disorders, mental retardation, substance dependence (abuse), etc.; Has active suicidal ideation (≥ 4 points on item 10 of the MADRS);
* Risk of serious injury to self or others;
* History of serious physical illness or disease that may affect the central nervous system;
* Risk of neurologic disorders or seizures, such as previous craniosynostosis, cranial trauma, abnormal electroencephalograms, magnetic resonance evidence of structural abnormalities of the brain, or family history of epilepsy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale（MADRS） | * "Baseline" * "Day 5" * "2 weeks after the end of temporal interference stimulation" * "4 weeks after the end of temporal interference stimulation"
  Montgomery-Asberg Depression Rating Scale (MADRS) is used to reflect the effect of antidepressant treatment and monitor the change of patients' condition. The scale is a separate scale, and the score should be based on clinical interviews. The symptoms should be asked from broad to detailed, so as to accurately score the severity. The rater must determine whether the score is on the defined score values (0,2,4,6) or between these scores (1,3,5), according to clinical practice. MADRS has a minimum value of 0 and a maximum value of 60, with larger scores representing poorer results.

SECONDARY OUTCOMES:
Hamilton Depression Scale（HAMD-17) | * "Baseline" * "Day 5" * "2 weeks after the end of temporal interference stimulation" * "4 weeks after the end of temporal interference stimulation"
  The Hamilton Depression Scale（HAMD-17) was used to assess the extent of the patient's depressive episodes, with higher scores representing more severe depression, and this scale was used to monitor the patient's improvement in depression before and after treatment. HAMD-17 has a minimum value of 0 and a maximum value of 52, with larger scores representing poorer results.
Hamilton Anxiety Scale（HAMA） | * "Baseline" * "Day 5" * "2 weeks after the end of temporal interference stimulation" * "4 weeks after the end of temporal interference stimulation"
  The Hamilton Anxiety Scale is primarily used for the assessment of anxiety levels, and has 14 items, each of which has a 0-4 scale, with anxiety possible above a score of 7. HAMA has a minimum value of 0 and a maximum value of 56, with larger scores representing poorer results. The higher the score, the more severe the anxiety.
Young Mania Rating Scale（YMRS） | * "Baseline" * "Day 5" * "2 weeks after the end of temporal interference stimulation" * "4 weeks after the end of temporal interference stimulation"
  The Young Mania Rating Scale is mainly used to assess the manic symptoms of the subjects before and after the treatment, there are 11 items, each symptom has a working scale, divided into 5 levels, the level score of each item is different, most of them are 0-4, in which the 5th, 6th, 8th and 9th items are scored as 0, 2, 4, 6, 8, and the higher the total score of the subject the more serious the degree of mania. YMRS has a minimum value of 0 and a maximum value of 60, with larger scores representing poorer results.
Snaith-Hamilton Pleasure Scale（SHAPS） | * "Baseline" * "Day 5" * "1 week after the end of temporal interference stimulation" * "2 weeks after the end of temporal interference stimulation" * "4 weeks after the end of temporal interference stimulation"
  The Snaith-Hamilton Pleasure Scale is a self-report scale that assesses the degree of the subject's pleasure deficit; the higher the score, the more severe their pleasure deficit. The scale was used to assess the degree of improvement in the patients' pleasure deficit before and after treatment. The minimum value of SHAPS is 14 and the maximum value is 56, with larger scores representing poorer results.
Temporal Experience of Pleasure Scale (TEPS) | * "Baseline" * "Day 5" * "1 week after the end of temporal interference stimulation" * "2 weeks after the end of temporal interference stimulation" * "4 weeks after the end of temporal interference stimulation"
  The Temporal Experience of Pleasure Scale (TEPS) is a self-report scale that assesses an individual's anticipation and experience of future pleasure, with higher scores suggesting a stronger experience of pleasure. The scale was used to evaluate the degree of improvement of pleasure deficit before and after treatment. The TEPS scale has a maximum value of 120 and a minimum value of 20. Lower scores indicate higher levels of pleasure deficit, while higher scores indicate higher levels of pleasure experience.
Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR) | * "Baseline" * "Day 1-5" * "1 week after the end of temporal interference stimulation" * "2 weeks after the end of temporal interference stimulation" * "4 weeks after the end of temporal interference stimulation"
  The Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR) is a self-report scale with 16 items that is primarily used to assess patients' depressive symptoms. The QIDS-SR scale has a minimum value of 0 and a maximum value of 27, with higher scores indicating poorer results.
Self-Rating Depression Scale (SDS) | * "Baseline" * "Day 5" * "1 week after the end of temporal interference stimulation" * "2 weeks after the end of temporal interference stimulation" * "4 weeks after the end of temporal interference stimulation"
  The Self-Rating Depression Scale (SDS), a 20-item, 4-point scale, is used to assess the severity of an individual's depressive symptoms. The SDS scale has a maximum value of 100 and a minimum value of 25, with larger scores representing poorer results.
Self-Rating Anxiety Scale (SAS) | * "Baseline" * "Day 5" * "1 week after the end of temporal interference stimulation" * "2 weeks after the end of temporal interference stimulation" * "4 weeks after the end of temporal interference stimulation"
  The Self-Rating Anxiety Scale (SAS) contains 20 items reflecting subjective feelings of anxiety, and each item is rated on a four-point scale according to the frequency of the symptom, with 15 positive ratings and 5 negative ratings (marked with an asterisk *), which allows the scale to rate the severity of anxiety symptoms and their change in treatment. The SAS scale has a maximum value of 100 and a minimum value of 25, with larger scores representing poorer results.
THINC-integrated tool (THINC-it) | * "Baseline" * "Day 5" * "2 weeks after the end of temporal interference stimulation" * "4 weeks after the end of temporal interference stimulation"
  THINC-it tool for assessing cognitive function changes in patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China